CLINICAL TRIAL: NCT03129035
Title: Bilateral Internal Iliac Artery Ligation Before Cesarean Hysterectomy : A Randomized Controlled Trial
Brief Title: Bilateral Internal Iliac Artery Ligation Before Cesarean Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2017-04-20; First posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- internal iliac artery ligation (Active Comparator): women undergo bilateral internal iliac artery ligation after fetal extraction and before proceeding in cesarean hysterectomy
  Interventions: Procedure: Cesarean hystrectomy; Procedure: Internal iliac artery ligation
- No internal iliac artery ligation (Active Comparator): Women undergo cesarean hysterectomy after fetal extraction
  Interventions: Procedure: Cesarean hystrectomy

INTERVENTIONS:
Procedure: Cesarean hystrectomy — Upper segment cesarean section followed by fetal extraction and cesarean hystrectomy started without any attempts of placental removal
Procedure: Internal iliac artery ligation — The retroperitoneal space was entered at the level of common iliac bifurcation and followed to the point of division into the external and internal iliac arteries. The ureter was retracted medially by gentle finger dissection, revealing the retroperitoneal anatomy. The fat and loose connective tissue around the IIA and vein were removed and a right-angle clamp was passed beneath the IIA from the lateral to the medial side approximately 4 cm distal to its origin. Using an absorbable suture, the IIA was ligated doubly in all cases . Pulsations of the external iliac and femoral arteries were identified after internal iliac ligation. The procedure was then repeated on the other side
  Arms: internal iliac artery ligation

SUMMARY:
All women with placenta accreta will be managed by upper segment cesarean section followed by cesarean hysterectomy without attempts of placental removal.

Women were randomized to either bilateral internal iliac artery ligation before hysterectomy and after fetal extraction or no additional intervention

DETAILED DESCRIPTION:
All women with placenta accreta will be managed by upper segment cesarean section followed by cesarean hysterectomy without attempts of placental removal.

Women were randomized to either bilateral internal iliac artery ligation before hysterectomy and after fetal extraction or no additional intervention.

Midline incision in the all patients is preferred. The retroperitoneal space was entered at the level of common iliac bifurcation and followed to the point of division into the external and internal iliac arteries. The ureter was retracted medially by gentle finger dissection, revealing the retroperitoneal anatomy. The fat and loose connective tissue around the IIA and vein were removed and a right-angle clamp was passed beneath the IIA from the lateral to the medial side approximately 4 cm distal to its origin.

Using an absorbable suture, the IIA was ligated doubly in all cases . Pulsations of the external iliac and femoral arteries were identified after internal iliac ligation. The procedure was then repeated on the other side.

ELIGIBILITY:
Inclusion Criteria:

* women with suspected placenta accreta
* Scarred uterus
* Approving hysterectomy

Exclusion Criteria:

* Women needed conservative surgery
* women with coagulopathy or bleeding disorders

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants needed blood transfusion | within 24 hours from surgery
  number of cases in each group who needed blood transfusion whether intraoperative or within 24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes